CLINICAL TRIAL: NCT07141004
Title: A Phase-IV, Multicenter, Non-Comparative, Open-Label Study Evaluating the Safety and Efficacy of Guselkumab Administered Subcutaneously in the Treatment of Indian Patients With Psoriatic Arthritis
Brief Title: A Study of Guselkumab Administered Subcutaneously in Treatment of Indian Participants With Psoriatic Arthritis (PsA)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNTO1959PSA4018; CNTO1959PSA4018 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2025-08-21; First posted 2025-08-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — guselkumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guselkumab (Experimental): Participants will receive subcutaneous injections of guselkumab at Weeks 0, 4, 12, and 20.
  Interventions: Drug: Guselkumab

INTERVENTIONS:
Drug: Guselkumab — Guselkumab will be administered as subcutaneous injection.
  Other Names: TREMFYA

SUMMARY:
The purpose of this study is to evaluate the safety and how well guselkumab treatment works (efficacy) in participants with psoriatic arthritis (PsA; a chronic, autoimmune form of arthritis that causes joint inflammation) who had inadequate response to standard therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have definite diagnosis of active psoriatic arthritis (PsA) (according to the ClASsification criteria for Psoriatic Arthritis [CASPAR]) prior to the first administration of study drug and have at least 1 of the PsA subsets: distal interphalangeal joint arthritis, polyarticular arthritis with the absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Participants who are negative for rheumatoid factors
* Participants having inadequate response (defined by presence of active arthritis [presence of any swollen or any tender joint]) to standard therapies for 3 months at the highest recommended dose (e.g., conventional disease-modifying antirheumatic drugs [DMARDs] including methotrexate, apremilast, or nonsteroidal anti-inflammatory drugs [NSAIDs]), including biologics naïve patient or have failed, or were intolerant to one or more biological treatments [anti-TNF/IL-17i]
* Participants are considered eligible per the following Tuberculosis (TB) screening criteria:

  1. Have no history of TB prior to screening AND
  2. Have no signs or symptoms suggestive of active TB upon medical history and/or physical examination AND
  3. Have had no recent close contact with a person with active TB, or if there has been such contact, will be referred to a physician specializing in TB to undergo additional evaluation and, if warranted, receive appropriate treatment for latent TB prior to or simultaneously with the first administration of study drug AND
  4. Within 6 weeks prior to the first administration of study drug, have a negative QuantiFERON- TB Gold and a negative tuberculin skin test result, OR have a newly identified positive QuantiFERON-TB Gold or tuberculin skin test result during screening in which active TB has been ruled out and for which appropriate treatment for latent TB has been initiated either prior to or simultaneously with the first administration of study drug AND
  5. Have a chest radiograph (both posterior-anterior and lateral views), taken within 3 months prior to the first administration of study drug and read by a qualified radiologist, with no evidence of current active TB or old inactive TB
* Medically stable on the basis of physical examination, medical history, vital signs, and 12-lead ECG
* A woman of childbearing potential must have a negative highly sensitive serum beta-hCG at screening visit

Exclusion Criteria:

* History of latent or active granulomatous infection prior to screening
* Have a known clinically significant hypersensitivity to guselkumab or to any of the excipients
* Have had a serious infection, or have been hospitalized for an infection, or have been treated with intravenous (IV) antibiotics for an infection within 2 months prior to first administration of study intervention
* Has any known malignancy or has a history of malignancy, or a history of lymphoproliferative disease
* Have received, or are expected to receive, any live virus or bacterial vaccination within 3 months before the first administration of study intervention, during the study, or within 6 months after the last administration of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-08-12 (Actual); Primary Completion 2027-06-05 (Estimated); Study Completion 2027-09-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 32 weeks
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants With Serious Adverse Events (SAEs) | Up to 32 weeks
  A SAE is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a suspected transmission of any infectious agent via a medicinal product; is medically important.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieve an American College of Rheumatology (ACR) 20 Response at Week 12 | Week 12
  ACR 20 Response is defined as greater than or equal to (>=) 20 percent (%) improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=20 percent (%) improvement from baseline in 3 of following 5 assessments: 1) participant's assessment of pain using Visual Analog Scale (VAS; 0-100 millimeter [mm], 0 mm=no pain and 100 mm=worst possible pain), 2) participant's global assessment of disease activity by VAS scale range: 0 mm= very well to 100 mm= very poor, 3) physician's global assessment of disease activity using VAS (scale ranges from 0 = no arthritis to 100 = extremely active arthritis), 4) participant's assessment of physical function measured by Health Assessment Questionnaire-disability Index (HAQ-DI). The derived HAQ-DI ranges from 0 indicating no difficulty to 3 indicating inability to perform a task in that area, and 5) C-reactive protein (CRP) and erythrocyte sedimentation rate (ESR).
Percentage of Participants Who Achieve an ACR 20 Response at Week 24 | Week 24
  ACR 20 Response is defined as >= 20% improvement from baseline in both swollen joint count (66 joints) and tender joint count (68 joints) and >=20% improvement from baseline in 3 of following 5 assessments: 1) participant's assessment of pain using VAS (0-100 mm, 0 mm=no pain and 100 mm=worst possible pain), 2) participant's global assessment of disease activity by using VAS (scale range: 0 mm= very well to 100 mm= very poor), 3) physician's global assessment of disease activity using VAS (scale ranges from 0 = no arthritis to 100 = extremely active arthritis), 4) participant's assessment of physical function measured by HAQ-DI. The derived HAQ-DI ranges from 0 indicating no difficulty to 3 indicating inability to perform a task in that area, and 5) CRP and ESR.
Change From Baseline in Analytic Marker of Inflammation (CRP Levels) at Weeks 12 and 24 | Baseline, Weeks 12 and 24
  CRP levels that is the analytic markers of inflammation will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- India (8):
  - Cims Hospital, Ahmedabad
  - Chennai Meenakshi Multispeciality Hospital, Chennai
  - Nizams Institute of Medical Sciences, Hyderabad
  - P. D. Hinduja National Hospital and Research Center, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - All India Institute of Medical Sciences, Patna
  - Jehangir Clinical Development Centre, Pune

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency